CLINICAL TRIAL: NCT06928987
Title: Evaluation of the Efficiency of Touch Massage on the Quality of Life at Work of Nursing Staff Working in a Cancer Center
Brief Title: Evaluation of the Efficiency of Touch Massage on the Quality of Life at Work of Nursing Staff Working in a Cancer Center. (Pause "Toucher Massage (TM)")
Acronym: PauseTM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICO-2023-22
Record Dates: First submitted 2024-11-05; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Quality of Life at Work; Paramedical Professionals; Touch Massage; Cancer Center
Keywords: burnout; stress; anxiety; affect; musculoskeletal disorders; well-being
MeSH Terms: conditions — Burnout, Psychological; Anxiety Disorders; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Touch massage (Experimental): Participants receive 6 Touch Massage sessions, given once a week for 6 weeks by one of the Touch Massage practitioners
  Interventions: Other: Touch Massage
- Without Touch massage (No Intervention): Participants will not receive any Touch Massage sessions for the duration of the study.

INTERVENTIONS:
Other: Touch Massage — The practitioner performs the touch-massage for 15 minutes on clothed personnel in a seated position on an ergonomic massage chair. The massage focuses on the back, neck and arm areas. It's a precise, technical sequence of pressure, stretching and sweeping movements that follows the following pattern:
  * Basic anti-stress maneuvers to relieve tension,
  * Relaxation of the upper torso with weightless movements to loosen shoulders and arms,
  * Stretching,
  * Redynamization through rapid friction on the back.
  Burnout, anxiety, affect, and musculoskeletal disorders (MSDs) will be assessed in participants using the following questionnaires at different times of the study.
  Arms: Touch massage

SUMMARY:
The goal of this clinical trial is to scientifically confirming the common perception that Touch-Massage (TM) breaks have a beneficial effect on the daily life of paramedics, both psychologically and physically.

The main question[s] it aims to answer [is/are]:

* Evaluating the efficacy of TM on burnout
* Evaluating the efficacy of TM on anxiety
* Evaluating the efficacy of TM on affect
* Evaluating the efficacy of TM on musculoskeletal disorders Researchers will compare 2 groups : Control group of paramedics who do not have the benefit of TM breaks and an experimental group of paramedics taking TM break.

Participants in the experimental group received one 15-minute TM session per week for 6 weeks and burnout, anxiety, affect, and musculoskeletal disorders (MSDs) will be assessed in participants using questionnaires at different times of the study. Participants in the control group complete only the same questionnaires at the same times as the experimental group.

Participants in the 2 arms are reviewed at 3 and 6 months to complete the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Nurses or nursing assistant working in the Institut de Cancérologie de l'Ouest's (ICO) medical oncology, surgical oncology, day clinic or early phase unit.
* Employees who have worked at the ICO for at least 9 months.

Exclusion Criteria:

* Employees who have had more than one touch/massage session at the ICO in the last 6 months.
* Pregnant for more than 4 months (declarative)
* Employees who have undergone osteo-articular surgery within the last 3 months.
* Employees with a pre-inclusion MBI score indicating high burnout (emotional exhaustion score >30 and depersonalisation score >12 and personal accomplishment score <33).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Burn out | At enrolment and at the end of the 6th session of touch massage (1 session per week for 6 weeks)
  Burnout is assessed using the Maslach Burnout Inventory (MBI) questionnaire, which consists of 3 scales (emotional exhaustion, depersonalisation and personal accomplishment).
  This score is obtained by adding items 1, 2, 3, 6, 8, 13, 14, 16 and 20, each of which is rated on a 7-point Likert scale (from 0=never to 6=every day).
  * Total < 17: low burnout
  * Total between 18 and 29: moderate burnout
  * Total > 30: high burnout

SECONDARY OUTCOMES:
Anxiety | At enrolment, at the end of the 6th session of touch massage (1 session per week for 6 weeks) and 6 months after randomisation
  Anxiety will be assessed using the State Trait Anxiety Inventory (STAI TRAIT) questionnaire. The questionnaire consists of 20 items that participants answer on a 4-point scale. Scores range from 20 to 80, with higher scores indicating greater anxiety.
Affect | At enrolment, at the end of the 6th session of touch massage (1 session per week for 6 weeks), at 3 and 6 months after randomisation
  Affect will be assessed using the Positive And Negative Affectivity Scale (PANAS). The questionnaire consists of 10 items assessing positive and negative affectivity. For each item, the participant responds on an ordered scale of 1 to 5, making it possible to calculate a score ranging from 10 to 50 for each dimension.
Musculoskeletal disorders | At enrolment, at the end of the 6th session of touch massage (1 session per week for 6 weeks), at 3 and 6 months after randomisation
  Musculoskeletal disorders will be assessed using the Nordic Musculoskeletal Questionnaire (NMQ). This questionnaire is used to record problems such as pain, discomfort and numbness in different parts of the body over the past 12 months and also over the past 7 days. It can also be used to assess the intensity of the problem at the time the questionnaire is completed.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancérologie de l'Ouest, Saint-Herblain, France